CLINICAL TRIAL: NCT07292389
Title: Examining Valence-based Effects in Self-monitoring Feedback Messages, in the Development of a Novel Semi-automated Self-monitoring Feedback System for Obesity Treatment
Brief Title: Examining Valence-based Effects in Self-Monitoring Feedback Messages
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: University of Florida (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Rebecca A. Krukowski, Principal Investigator, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB302281
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Obesity & Overweight; Obesity (Disorder)
Keywords: weight loss; self-monitoring; smartphone app; lifestyle intervention; digital health; physical activity; dietary change; e-scale; wearables; activity monitor; behavior change; self-monitor activity
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Motor Activity

STUDY DESIGN:
Intervention Model Description: Micro-randomized Factorial. One of two conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self Monitoring Feedback (Experimental): Participants in this study will complete a 60-minute "Weight Loss 101" session and use study-provided tools to record their daily food intake, physical activity, and weight. After a one-week run-in period, they will begin receiving weekly feedback messages. The content and emphasis of these messages will differ between 2 conditions: positive reinforcement vs. positive reinforcement + areas for change.
  Interventions: Behavioral: Positive Reinforcement; Behavioral: Positive Reinforcement + Areas for Change

INTERVENTIONS:
Behavioral: Positive Reinforcement — Feedback composed by a study interventionist that focuses exclusively on positively reinforcing the participant's progress toward achieving their goals.
Behavioral: Positive Reinforcement + Areas for Change — Feedback provided by a study interventionist that combines positive reinforcement of the participant's progress with constructive guidance on areas for improvement to support successful goal attainment.

SUMMARY:
The purpose of this research study is to learn how to identify the most effective ways to provide weekly feedback on participants' progress toward intervention goals during a weight loss program.

DETAILED DESCRIPTION:
This micro-randomized factorial trial is designed to provide information about how to optimize self-monitoring feedback within a behavioral weight management intervention. All participants will attend a "Weight Loss 101" session that covers foundational weight loss education and behavioral skills training. During this session, they will also learn how to use study-provided tools to track their dietary intake, physical activity, and weight.

Each weekly feedback message will be composed by a trained interventionist. Participants will be randomized each week to one of the two conditions to examine how the tone and composition of feedback messages impact participant behaviors and weight loss.

The main questions that this study aims to answer are:

* How does the composition of supportive feedback and ideas for potential changes in dietary or physical activity behaviors impact weight loss.
* How is this feedback affected by individual or contextual factors?

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* BMI greater than or equal to 25.0 kg/m2
* Weight less than or equal to 175 kg (due to scale limit)
* Own a smartphone compatible with Fitbit (e.g., an Apple iPhone running iOS 16.4 or higher or Android smartphone running Android 11 or higher) with a cellular and data plan

Exclusion Criteria:

* Weight greater than 175 kg (due to a weight limit of the study-provided scale)
* Smartphone device owned deemed incompatible with the Fitbit App
* History of bariatric surgery or plans to obtain bariatric surgery during the study period
* Current use of weight loss medications, or use of weight loss medications in the 6 months prior to initial pre-screening
* Currently participating in a weight-loss program
* Weight loss of greater than or equal to 10 lbs in the 6 months prior to initial pre-screening
* Physical limitations that prevent walking at a brisk pace for at least 10 minutes without stopping
* Use of a pacemaker or other implanted medical device
* Currently pregnant
* Currently breastfeeding
* Less than 1-year post-partum
* Plans to become pregnant within the study period
* Lack of written confirmation that the potential participant has discussed study participation with their physician if they have been diagnosed with diabetes, hypertension, or has have a history of coronary heart disease
* One or more study participants living in the household (enrollment limited to one participant per household)
* Medical conditions that contraindicate weight loss or prevent completion of the study (e.g., current diagnosis of cancer or terminal illness, dementia, etc.)
* Recent (in the past 6 months) changes in medications that affect weight
* Self-reported eating disorder within past 5 years
* Unable to complete the 17-week study (due to plans to relocate during the study period, etc.)
* Unable or unwilling to provide informed consent
* Unable to read English at the 5th grade level
* Unwilling to accept random assignment
* Unable or unwilling to download the study smartphone application, wear the physical activity monitor, or use the study e-scale
* Failure to complete baseline assessment measures
* Failure to complete at least 4 out of 6 days of self-monitoring dietary and weight self-monitoring during the behavioral run-in period
* Any other condition(s) which, in the opinion of the Principal Investigator, would adversely affect participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Weight change | 7 days
  Mixed-effects models will be used to investigate the impact of each feedback condition on our primary outcome of weight change. Fitted model estimates will be used to calculate the slope of weight change from day 1 (the day a feedback message is delivered) through day 7 of each week. Positive slopes indicate weight gain, while negative slopes indicate weight loss.

SECONDARY OUTCOMES:
Frequency of self-monitoring weight | 7 days
  Frequency of self-monitoring weight will be defined as the number of days (0-7) in the week following a feedback message (from day 1, the day that a feedback message is received, to day 7) in which the participant records a valid (non-outlier) e-scale weight.
Frequency of self-monitoring dietary intake | 7 days
  A valid "day" of dietary self-monitoring will be defined as ≥ 800 kcal recorded, consistent with prior research. Frequency is calculated as the number of valid days (0-7) recorded the week after a feedback message is delivered (from day 1, the day that a feedback message is received, to day 7).
Total caloric intake | 7 days
  Total caloric intake will be calculated by summing calories consumed during the week following a feedback message is received (from day 1, the day that a feedback message is received, to day 7)
Calorie goal attainment | 7 days
  Calorie goal attainment for each day during the week after a feedback message is received (from day 1, the day a feedback message is received, to day 7). Calorie goal attainment will be calculated as [TOTAL KCAL INTAKE FOR THE DAY] - [CALORIE GOAL]. Daily difference scores for the 7 days will be averaged across the week to determine overall adherence to the caloric intake goal.
Frequency of self-monitoring physical activity | 7 days
  Frequency of self-monitoring physical activity will be defined as the number of "valid" days (0-7) of Fitbit use the week after a feedback message is received (from day 1, the day that a feedback message is received, to day 7).
Physical activity minutes | 7 days
  Total minutes of physical activity will be calculated by summing each days' total "active zone minutes" during the week after a feedback message is delivered (from day 1, the day that a feedback message is received, to day 7)
Physical activity goal attainment | 7 days
  Physical activity goal attainment for each day of the week after a feedback message is received (from day 1, the day that a feedback message is received, to day 7) will be calculated as [TOTAL PHYSICAL ACTIVITY MINUTES] - [PHYSICAL ACTIVITY GOAL]. Daily difference scores will be averaged over the week to assess overall adherence to the physical activity goal during that study week.

CONTACTS AND LOCATIONS:
Overall Officials: Becca Krukowski, Ph.D., Principal Investigator — University of Virginia

IPD SHARING:
Plan to Share IPD: Yes
Individual-level participant data will be de-identified and made available at the time of publication of peer-reviewed manuscript(s) based on the data. Study data will be shared via the Zenodo data repository at https://zenodo.org/. Analytic code will be made publicly available via Supplementary files for any publications and/or via Zenodo through a Zenodo-GitHub link. Study protocol, informed consent form, statistical analysis plan will also be available to be shared via clinicaltrials.gov.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified, individual-level participant data will be made available at the time of publication of peer-reviewed manuscript(s) based on the data.
Access Criteria: Data will be made available via the Zenodo data repository (https://zenodo.org).
URL: https://zenodo.org/